CLINICAL TRIAL: NCT02896816
Title: EMG Modules as a Novel Biomarker of Basal Ganglia Plasticity in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No more funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2015-P-002526
Record Dates: First submitted 2016-06-29; First posted 2016-09-12 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Parkinson
Keywords: Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's subjects (Experimental): The participants with Parkinson's disease should have symptoms only on one side of the body, and they should not be taking any dopamine replacement medication such as levodopa or dopamine agonists.
  Surface EMG, MRI and PET scan will be performed at baseline.
  Interventions: Other: Surface EMG, MRI and PET Scan
- Control subjects (Active Comparator): Participants not affected by neurological disorders. Surface EMG will be performed at baseline.
  Interventions: Other: Surface EMG

INTERVENTIONS:
Other: Surface EMG, MRI and PET Scan — It will consist of two assessment sessions; one where muscle activity of the arms as well as movement characteristics will be assessed during a reaching task; and another where muscle activity of the legs and movement characteristics will be assessed while walking on a treadmill. Clinical evaluations will also be performed. In addition, individuals with Parkinson's disease will undergo brain scans at Massachusetts General Hospital to examine whether there are any relationships between muscle activity and brain function.
  Arms: Parkinson's subjects
Other: Surface EMG — It will consist of two assessment sessions; one where muscle activity of the arms as well as movement characteristics will be assessed during a reaching task; and another where muscle activity of the legs and movement characteristics will be assessed while walking on a treadmill. Clinical evaluations will also be performed.
  Arms: Control subjects

SUMMARY:
Study Purpose:

Parkinson's disease leads to severally impaired motor control. The purpose of this study is to better understand and analyze the characteristics of arm muscle activity while doing some reaching tasks and of leg muscles while walking. This will allow the investigators to improve understanding of the mechanisms underlying the motor impairments in Parkinson's disease.

DETAILED DESCRIPTION:
More details:

A total of 20 participants with Parkinson's disease and 20 age- and gender-matched healthy controls will be included in this study. The participants with Parkinson's disease should have symptoms only on one side of the body, and they should not be taking any dopamine replacement medication such as levodopa or dopamine agonists. The study will take place at the Motion Analysis Laboratory of Spaulding Rehabilitation Hospital in Charlestown, Massachusetts. It will consist of two assessment sessions; one where muscle activity of the arms as well as movement characteristics will be assessed during a reaching task; and another where muscle activity of the legs and movement characteristics will be assessed while walking on a treadmill. Clinical evaluations will also be performed. In addition, individuals with Parkinson's disease will undergo brain scans at Massachusetts General Hospital to examine whether there are any relationships between muscle activity and brain function.

ELIGIBILITY:
Inclusion Criteria for Parkinson's volunteers:

1. Male and female, age 18-80
2. Motor symptoms only on one side of the body
3. No use of dopaminergic replacement therapy or other medication related to PD

Exclusion Criteria for Parkinson's volunteers:

1. Cognitive impairments that may interfere with understanding instructions as needed during the performance of the study (MMSE<23)
2. Subjects who are unable to perform arm reaching movements
3. Self-report of any condition that could affect walking
4. No fractures or skin lesions in the upper or lower limbs
5. Infectious diseases requiring contact precautions
6. Subjects with contraindications to MRI cannot participate (i.e., implanted metal including pacemakers, cerebral spinal fluid shunts, aneurysm clips, artificial heart valves, ear implants or metal/foreign objects in the eyes and those with a history of claustrophobia)
7. Pregnancy: If the possibility of pregnancy of a female participant cannot be excluded by: 1) surgical history (e.g., tubal ligation or hysterectomy) or 2) post menopausal status with a minimum of 1 year without menses, then a pregnancy test by stat serum testing must be performed on site the morning of any PET visit and the negative result is required prior to the administration or any radiopharmaceutical
8. Substance abuse within the past 2 years as it may alter neurotransmitter function
9. Active hematological, renal, pulmonary, endocrine or hepatic disorders
10. Evidence of cortical infarcts or strategically placed lacunar infarct (e.g. dorsal medial nucleus of thalamus)
11. Active cancer, metabolic encephalopathy, infection
12. Active cardiovascular disease, stroke, congestive heart failure
13. Diagnosis of MCI or dementia

Inclusion criteria for healthy volunteers:

1. Male and female, age 18-80
2. Age and gender-matched to PD patients
3. No use of dopaminergic replacement therapy or other medication related to PD

Exclusion criteria for healthy volunteers:

1. Cognitive impairments that may interfere with understanding instructions as needed during the performance of the study (MMSE<23)
2. Subjects who are unable to perform arm reaching movements
3. Self-report of any condition that could affect walking
4. No fractures or skin lesions in the upper or lower limbs
5. Infectious diseases requiring contact precautions
6. Diagnosis of MCI or dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Surface electromyography recording | Baseline
  Surface EMG upper and lower extremities

SECONDARY OUTCOMES:
Structural MRI | Baseline
  T1 and T2 structural MRI will be performed.
Functional MRI | Baseline
  Resting state and task functional MRI will be performed to obtain BOLD signals.
Diffusion weighted imaging | Baseline
  Diffusion weighted imaging will be performed to obtain connectivity measures.
Altropane PET scan | Baseline
  Altropane PET scan will be performed to assess dopamine transport

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No